CLINICAL TRIAL: NCT06768034
Title: A Pilot Pragmatic Randomized Controlled Trial Evaluating Secondary Cardiovascular Prevention Therapies in Patients Who Had a Myocardial Injury After Noncardiac Surgery to Prevent Major Cardiovascular Events
Brief Title: SecondarY Prevention and MaNagement of Myocardial Injury AftER Noncardiac SurGerY (SYNERGY) Pilot Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Emmanuelle Duceppe MD PhD, Scientist, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-12117
Record Dates: First submitted 2024-12-20; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Injury After Noncardiac Surgery (MINS)
Keywords: Noncardiac surgery; Secondary cardiovascular prevention; Randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Patients who had myocardial injury after noncardiac surgery are assigned to receive usual care.
- Systematic referral for secondary cardiovascular prevention (Active Comparator): Systematic referral to an internist within 6 weeks after myocardial injury after noncardiac surgery for implementation of secondary cardiovascular prevention strategies, individualized the patient's risk factors.
  Interventions: Procedure: Intervention Group

INTERVENTIONS:
Procedure: Intervention Group — Patients being referred to an internist or cardiologist after myocardial injury after noncardiac surgery
  Arms: Systematic referral for secondary cardiovascular prevention

SUMMARY:
Cardiac complications, particularly myocardial injury after noncardiac surgery (MINS), significantly contribute to 30-day mortality, affecting about 1 in 10 patients after noncardiac surgery. Despite its prevalence and serious implications, there is no consensus on managing myocardial injury after noncardiac surgery in clinical practice. Interventions commonly used for cardiovascular prevention in patients who had a heart attack outside of a surgery context could also be beneficial in patient with MINS. This pilot study trial aims to gather feasibility data, such as recruitment rates and intervention adherence that will guide on the design and inform on sample size of a future study with large pragmatic randomized controlled trial on the impact of systematic referral for secondary cardiovascular prevention on outcomes in patients who had a MINS.

DETAILED DESCRIPTION:
The SYNERGY study is a pilot randomized controlled trial with 100 patients who had myocardial injury after noncardiac surgery (MINS). Patients are assigned to either a control group receiving usual care or an intervention group that receives referral to a specialist for implementations of interventions on secondary cardiovascular prevention. Secondary cardiovascular prevention will be individualized to the patient's risk factors and may include antiplatelet agents, cholesterol-lowering treatment, blood pressure-lowering medication, as well as counselling on healthy lifestyle choices on diet and exercise, including, if applicable, optimization of diabetes treatment and help in quitting smoking.

At six months, follow-up will assess clinical cardiovascular outcomes, medication adherence, smoking status, adherence to a Mediterranean diet and physical activity.

Key feasibility metrics include recruitment rate, intervention adherence, crossover in the control group, and changes physical activity and dietary pattern. This study aims to address untreated myocardial injury after noncardiac surgery by collecting feasibility data to inform on the design of a future large randomized clinical trials on secondary cardiovascular prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Have undergone noncardiac surgery,
2. Had a myocardial injury after noncardiac surgery with a presumed ischemic mechanism and without an overt nonischemic precipitating etiology (e.g., sepsis)
3. Provide written informed consent to participate in the SYNERGY pilot trial.

Exclusion Criteria:

1. already on 2 of 3 secondary cardiovascular prevention medications (i.e., antiplatelet, statin, and/or angiotensin-converting enzyme inhibitor (ACEI)/angiotensin II receptor blocker (ARB)
2. patients with contraindication to statins (i.e., decompensated or Child-Pugh C cirrhosis, acute liver failure, elevated AST/ALT greater than 2-fold the normal upper limit, previous demonstrated statin hypersensitivity, allergy, or statin-related myopathy);
3. patients with contraindication to antiplatelet therapy (i.e., active or recent <1-month peptic ulcer disease, esophageal or gastric variceal disease, history of intracranial or intraspinal hemorrhage, significant thrombocytopenia with platelet count <50 × 109/L),
4. patients with contraindication to ACEI and ARB therapy (i.e, hypersensitivity or allergy to ACEI or ARB);
5. Previously enrolled in the SYNERGY pilot trial,
6. Considered unreliable or unable to complete the trial procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Average recruitment rate | 12 months
  Average number of patients recruited per month. Feasibility is defined as average recruitment rate ≥3 patients/month/site as "trial feasible", between 1-2 patients/month/site as "potentially feasible with protocol modifications", and <1 patient/month/site as "unlikely feasible".
Proportion adherence to referral to specialized cardiovascular care in the intervention group | 6 months
  Defined as the proportion of patients allocated to the intervention group with referral to internal medicine or cardiology within 6 weeks of MINS. The adherence feasibility outcome is defined as follows: ≥70% as "trial feasible", between 40-69% "potentially feasible with protocol modifications", and <40% "unlikely feasible".
Proportion crossover to referral to specialized CV care in the control group | 6 months
  Defined as the proportion of patients allocated to the control group with referral to internal medicine or cardiology within 6 weeks of MINS. The crossover feasibility outcome is defined as follows: <30% as "trial feasible", between 30-49% "potentially feasible with protocol modifications", and >50% "unlikely feasible".

SECONDARY OUTCOMES:
Proportion of prescription of cardiovascular medications | 6 months
  Proportion of patients who are prescribed an antiplatelet, statin, and angiotensin-converting enzyme inhibitor (ACEI)/angiotensin II receptor blockers (ARB) (all three) at 6 months.
Proportion of patients on antiplatelet therapy | 6 months
  Proportion of patients who are prescribed an antiplatelet therapy.
Proportion of patients on statin therapy | 6 months
  Proportion of patients who are prescribed a statin.
Proportion of patients on angiotensin-converting enzyme inhibitor (ACEI)/angiotensin II receptor blocker (ARB) | 6 months
  Proportion of patients who are prescribed an angiotensin-converting enzyme inhibitor (ACEI)/angiotensin II receptor blocker (ARB).
Proportion consent of eligible patients | 12 months
  Proportion of eligible patients which consented to participate in the trial
Proportion of completeness to follow-up | 6 months
  Proportion of patients enrolled in the trial that completed the 6-month follow-up
Change in IPAQ score | 6 months
  Difference in physical activity score (i.e., the short form of the International Physical Activity Questionnaire (IPAQ-SF) score in metabolic equivalents (METs) minute per week) between baseline and 6 months, expressed as a continuous outcome, with higher values meaning a larger increase in physical activity level.
Change in MEDAS score | 6 months
  Difference between the Mediterranean Diet Adherence Screener (MEDAS) questionnaire score at baseline and 6 months (score between 0 and 14, with high score reflecting higher adherence).
Proportion of major cardiovascular events | 6 months
  Proportion of patients who experience any of the following composite of cardiovascular death, non-fatal cardiac arrest, myocardial infarction, stroke, heart failure, and coronary revascularization.
Proportion of cardiovascular death | 6 months
  Proportion of patients with a cardiovascular death is defined as any death with a cardiovascular cause and includes those deaths following a myocardial infarction, sudden cardiac arrest, stroke, cardiac revascularization procedure (i.e., percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery), and heart failure.
Proportion of myocardial infarction | 6 months
  Proportion of patients with a myocardial infarction as defined according to the Fourth Universal Definition of Myocardial Infarction.
Proportion of non-fatal cardiac arrest | 6 months
  Proportion of patients with a nonfatal cardiac arrest defined as successful resuscitation from either documented or presumed ventricular fibrillation, sustained ventricular tachycardia, asystole, or pulseless electrical activity requiring cardiopulmonary resuscitation, pharmacological therapy, or cardiac defibrillation.
Proportion of coronary revascularization | 6 months
  Proportion of patients with a cardiac revascularization procedures including percutaneous coronary intervention (PCI) and coronary arterial bypass grafting (CABG).
Proportion of stroke | 6 months
  Proportion of patients with a stroke defined as either:
  1. a new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting more than 24 hours or leading to death, OR
  2. a new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting less 24 hours with a positive neuroimaging consistent with a stroke.
Proportion of transient ischemic attack | 6 months
  Proportion of patients with a transient ischemic attack defined as rapidly developed and transient clinical signs of focal or global disturbance of cerebral function, lasting less than 24 hours, with either 1) direct weighted magnetic resonance findings of acute brain ischemic lesions, or 2) high risk neurologic features (i.e., lateralizing weakness and/or speech disruption lasting >5 min).
Proportion of heart failure | 6 months
  Proportion of patients with a diagnosis of heart fialure, as defined by (criteria A and B required):
  A. New or worsening symptoms due to heart failure (HF), including at least ONE of the following:
  1. Shortness of breath (dyspnea with exertion, dyspnea at rest, orthopnea, paroxysmal nocturnal dyspnea), 2. Decreased exercise tolerance, or 3. Fatigue.
  B. Signs of new or worsening HF, consisting of at least TWO physical examination findings OR one physical examination finding and at least ONE laboratory (i.e., natriuretic peptide elevation) or radiological imaging.
Proportion of all-cause mortality | 6 months
  Proportion of patients who died of any cause.
Proportion of new significant arrythmia | 6 months
  Proportion of patients with a new significant arrythmia defined as new supraventricular or ventricular arrythmia that results in angina, congestive heart failure, symptomatic hypotension, or that requires oral or intravenous treatment with a rate controlling drug, antiarrhythmic drug, electrical cardioversion, implantation of a pacemaker or implantable cardioverter defibrillator.
Proportion of major bleeding | 6 months
  Proportion of patients with a major bleeding defined according to the criteria of International Society on Thrombosis and Haemostasis (ISTH) as clinically overt bleeding which was fatal or associated with any of the following:
  1. a fall in hemoglobin level of 2 g/dL or more or documented transfusion of at least 2 units of packed red blood cells,
  2. involvement of a critical anatomical site (intracranial, spinal, ocular, pericardial, articular, intramuscular with compartment syndrome, retroperitoneal).
Proportion of clinically relevant non-major bleeding | 6 months
  Proportion of patients with a clinically relevant non-major bleeding defined as any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:
  1. requiring medical intervention by a healthcare professional
  2. leading to hospitalization or increased level of care
  3. prompting a face to face (i.e., not just a telephone or electronic communication) evaluation
Proprotion of kidney injury | 6 months
  Proportion of patients with a kidney Injury defined by the Acute Kidney Injury Network (AKIN) definition and classified according to the following stage:
  Stage 1: Serum creatinine increase ≥26.5 μmol/l or increase to 1.5-2.0-fold from baseline Stage 2: Serum creatinine increase >2.0-3.0-fold from baseline Stage 3: Serum creatinine increase >3.0-fold from baseline or serum creatinine ≥354 μmol/l with an acute increase of at least 44 μmol/l or need for new renal replacement therapy.
Proportion of liver injury | 6 months
  Proportion of patients with a liver injury defined by elevation of ALT and/or AST ≥3 times the upper limit of normal.
Proportion of rhabdomyolysis | 6 months
  Proportion of patients with a rhabdomyolysis defined as muscle symptoms with serum creatinine kinase ≥10 times the upper limit of normal.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Duceppe, MD PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No